CLINICAL TRIAL: NCT02825979
Title: Early Aggressive Invasive Intervention for Atrial Fibrillation
Acronym: EARLY-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jason Andrade (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); Medtronic (Industry); Baylis Medical Company (Industry)
Responsible Party: Sponsor-Investigator, Jason Andrade, MD, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-00617
Record Dates: First submitted 2016-05-18; First posted 2016-07-07 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sotalol; Flecainide; Propafenone; Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon-based PVI (Active Comparator): Sinus rhythm control via a pulmonary vein isolation (PVI) ("first-line") procedure utilizing the the Arctic Front Cryoballoon Procedure.
  Interventions: Procedure: Cryoballoon-based PVI
- Anti-Arrhythmic Drug Therapy (Active Comparator): Sinus rhythm control via the use of anti-arrhythmic drug (AAD) therapy ("first-line") based on local clinical practice, and according to guideline-suggested drug management for symptomatic patients with paroxysmal AF.
  Interventions: Drug: Anti-Arrhythmic Drug Therapy

INTERVENTIONS:
Procedure: Cryoballoon-based PVI — Patients randomized to first-line cryoballoon (CB) ablation will have the pulmonary vein isolation procedure performed according to standard clinical practice using the Arctic Front Cryoballoon ablation catheter. No anti-arrhythmic drugs will be prescribed in this arm.
  Arms: Cryoballoon-based PVI
Drug: Anti-Arrhythmic Drug Therapy — Antiarrhythmic drug therapy (Class I - flecainide, propafenone; Class III - sotalol, dronedarone) will prescribed and monitored based on local clinical practice, and according to guideline-suggested drug management for symptomatic patients with paroxysmal AF.
  Other Names: sotalol, flecainide, propafenone, dronedarone
  Arms: Anti-Arrhythmic Drug Therapy

SUMMARY:
The EARLY-AF study is centered on an evaluation of the impact of the early invasive management of Atrial Fibrillation. The primary goal of the study is to evaluate the clinical effectiveness of an early invasive approach. Specifically, the investigators are aiming to evaluate if PVI performed with the Arctic Front cryoballoon is superior to AAD as first-line therapy in preventing atrial arrhythmia recurrences (arrhythmia related symptoms, hospitalisations, and health care utilization) and health care utilisation at one year of follow-up. The aim of the extended follow-up phase of the trial (PROGRESSIVE-AF) is to evaluate if the initial treatment choice (ablation vs. pharmacotherapy) influences AF disease progression, as measured by continuous cardiac monitoring. The outcomes of interest are disease progression, quality of life, and healthcare utilisation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia seen in clinical practice, affecting approximately 1-2% of the overall population. Contemporary guidelines recommend AADs as the "first-line" therapy for the maintenance of sinus rhythm. However, these medications have only modest efficacy at maintaining sinus rhythm. Moreover, these agents are associated with significant non-cardiac side-effects, as well as the potential for pro-arrhythmia, heart failure, or organ toxicity. Conversely, the success rate of catheter ablation in maintaining sinus rhythm is universally superior to that of drug therapy when AADs have been ineffective, are contra-indicated, or cannot be tolerated. While catheter ablation has not been definitively proven to improve survival, it has been shown to be superior to AADs for the improvement of symptoms, exercise capacity, and quality of life.

Why consider early invasive intervention? Given the superiority of ablation over AAD therapy, it is postulated that early invasive intervention with catheter ablation offers an opportunity to halt the progressive pathophysiological and anatomical changes associated with AF. While catheter ablation has not been definitively proven to impact mortality in unselected patients, there are certain patient groups (e.g. younger patients, those with newly diagnosed AF, and those with heart failure) who may derive significant benefit from ablation. In addition, early invasive intervention may result in a significant reduction in overall health care utilitization.

The evidence supporting "first-line" catheter ablation (i.e. as an initial therapy prior to AAD) with radiofrequency (RF) energy is promising, but far from definitive. To date three key studies have been performed. The MANTRA-PAF Study and the RAAFT studies randomized patients to either first-line ablation or first-line AADs. Despite disparate ablation techniques, these studies collectively demonstrated an improved freedom from recurrent arrhythmia (37% reduction in AF recurrence vs. AAD therapy), an improved freedom from symptomatic AF (43% reduction in symptomatic AF vs. AAD therapy), and a reduction in the overall AF burden (50% reduction over AAD therapy). While the results of these previous studies suggest that ablation is more effective than AAD therapy as first-line treatment, a significant proportion of patients in the intervention group experienced arrhythmia recurrence.

STUDY DESIGN - The study is a multicenter prospective, open label randomized clinical trial with blinded adjudication of endpoints. Patients with untreated AF will be randomized in a 1:1 ratio to either first-line antiarrhythmic therapy or first-line AF ablation using cryothermal energy. Randomization will be performed with concealed allocation using permuted block randomization according to a computer-generated sequence (Dacima, Montreal, Canada). An independent, blinded statistician will generate the block randomization scheme. Outcomes will be adjudicated by personnel who are blinded to subjects' randomization status.

FUNDING The EARLY-AF study is funded by a peer-reviewed grant from the Cardiac Arrhythmia Network of Canada. In addition, the trial is supported by an unrestricted grant from Medtronic. The funding sources had no role in the design of this study and will not have any role during its execution, analyses, interpretation of the data, or decision to submit results.

STUDY POPULATION Patients aged ≥18 years with symptomatic, treatment naïve AF will be screened for eligibility. At least 1 episode of AF must be documented on 12-lead electrocardiogram (ECG), transtelephonic monitor (TTM), or Holter monitor within 24 months of randomization.

INTERVENTIONS All study participants will undergo the implantation of an ICM for the purpose of arrhythmia monitoring (Reveal LINQ™). The timing of the ICM implant will be no later than 24 hours after AAD initiation ("first-line" AAD group), and no later than 24 hours after the ablation procedure ("first-line" ablation group). ICM programmed parameters are summarized in Table 2. Participation in the trial is not possible without an ICM.

Patients randomized to AAD arm will start regular (daily) AAD therapy within 1 week of randomization. The use of AAD therapy will be based on local clinical practice, and according to guideline-suggested management for symptomatic patients with paroxysmal AF.4, 5 Suggested AAD titration and monitoring protocols are provided in Appendix E. During the titration phase, the ICM data will be reviewed by study personnel on a weekly basis, with AAD therapy progressively up-titrated to the maximum tolerated dose with a goal of complete AF suppression. In the event of clinical inefficacy or intolerable side effects, a change to a second or to a third AAD will be undertaken, insofar as the patient remains within the blanking period. Once the blanking period has ended, any further changes made to AAD therapy for recurrence of symptomatic or asymptomatic AF, atrial flutter, or atrial tachycardia would be considered a primary endpoint.

Patients randomized to catheter cryoablation will undergo the procedure within 2 months of randomization. Ablation may be performed under conscious sedation or general anesthesia, per local practice. The 28 mm cryoballoon catheter (Arctic Front Advance, Medtronic) will be advanced through the steerable sheath into the LA with a 20-mm small-diameter circular mapping catheter inserted in the central lumen of the CB and used as a guidewire. In exceptional circumstances the 23-mm cryoballoon may be used for PV diameters <20 mm and based on physician judgment. Cryoablation with a minimum ablation duration of 3 minutes will be utilized. Lesions that fail to isolate the vein within 60 seconds (if real-time PV potential monitoring is feasible) or achieve a temperature colder than minus 35oC after 60 seconds of ablation should be considered ineffectual and be terminated (except for common ostia). Thereafter the balloon and/or guidewire should be repositioned and a new lesion delivered. Once PVI has been achieved a single "bonus" application of 3 minutes will be delivered following the rewarming phase (to +20oC). Should the operator fail to isolate the PV (excluding common ostia) after a minimum of 3 attempted cryoballoon applications then focal ablation with the 8mm cryocatheter targeted to sites of LA-PV breakthrough will be permitted at operator discretion.

Post therapeutic intervention "Blanking period" In accordance with 2017 expert consensus statement for reporting outcomes in AF ablation trials, a blanking period of 3 months is incorporated for both groups.19 The rationale for the post-procedure blanking period is based on the observation that early recurrences of arrhythmias are common during the initial 3 month period post ablation, and is predicated on the assumption that not all early recurrences of atrial tachyarrhythmias (AF/AFL/AT) will lead to later recurrences and, as such, does not necessarily represent treatment failure. Correspondingly the 3-month "blanking period" in the AAD group will allow for drug titration and optimization. For this group the ICM data will be reviewed on a weekly basis to guide AAD titration during the blanking period.

Anticoagulation All patients will be systemically anticoagulated based on perceived stroke risk as per treatment guidelines and physician discretion. The decision to initiate oral anticoagulation will be made based on the risk of stroke as per the CCS algorithm. In patients <65 years of age and with a CHADS score of 0, aspirin alone or no specific antithrombotic therapy may be considered at treating physician discretion. For those >65 years of age, or with a CHADS score of 1 or more, OAC is strongly recommended. In the ablation group, all patients with a CHA2DS2-VASc ≥1 will remain anticoagulated with oral vitamin K antagonists (target INR between 2-3), low molecular weight heparin, or non-VKA oral anticoagulant medications for a minimum of 1 month prior to ablation and up to a minimum of 3 months post ablation. Thereafter, discontinuation of oral anticoagulation may be considered for patients <65 years of age and with a CHADS score of 0 (as above).

Minimization of Cross-Over All efforts will be undertaken to avoid patients switching from their randomized group to the alternate treatment strategy. However, patients with documented symptomatic arrhythmia recurrence may "change treatment strategy" (e.g. from AAD to ablation, or vice versa) if the arrhythmia event occurs outside the 90-day blanking period (i.e. constitutes a primary endpoint for the study). A "cross-over" will be defined if the patient changes treatment strategy within the blanking period or in the absence of documented AF.

For patients to "change treatment strategy" from the AAD group to the ablation group or vice versa, the symptomatic sustained arrhythmia recurrence must occur outside the blanking period. In the AAD group, recurrence must occur despite a therapeutic dose of AAD therapy (defined as flecainide >50 mg BID, sotalol >80 mg BID, or propafenone >150 mg BID, or dronedarone 400 mg BID). The recurrence should be of sufficient clinical severity to warrant the performance of an ablation procedure, as per standard clinical practice. Prior to permitting a patient to "change treatment strategy", an independent committee will review the rationale for change, the medication profile (to ensure adequate AAD dosing), and the arrhythmia episodes (which will have been independently adjudicated by the clinical events committee). Following this review, a change in treatment strategy may be permitted if the pre-specified criteria were met. If the patient is changing to ablation, the procedure should preferentially occur after the conclusion of the study follow-up but can occur sooner based on clinical necessity. The ablation procedure performed will preferably be a cryoballoon-based PVI (as outlined above).

ASSESSMENTS All patients will be followed for a minimum of 12 months after the index ablation procedure or medication initiation. This duration is based on the 2017 expert consensus statement for reporting outcomes in clinical trials of AF ablation, as well as the knowledge that most recurrences transpire during the first year after ablation.

Table 3 details the planned visits and procedures. For both groups, a one-week post treatment telephone call will occur followed by scheduled visits at 3, 6, and 12-months from index ablation procedure or medication initiation. A clinical evaluation and ECG will be performed at each of the scheduled clinical encounters. A specific patient interview will be conducted at each clinical visit to ascertain symptomatic AF. Information regarding disease specific HRQOL, generic HRQOL and an AF symptoms score will be assessed at each follow-up visit. In addition, information regarding health care resource use will be prospectively collected (emergent acute care visits, emergency department visits, hospitalizations, cardioversions, re-ablation, and planned/unplanned follow-up visits, and medication usage).

Automatic transmissions from the ICM will be obtained on a daily basis. In addition, we have instructed patients to identify symptomatic episodes through the use of the loop recorder's patient activator

Primary outcome - Time to first recurrence of symptomatic or asymptomatic AF, atrial flutter, or atrial tachycardia (AF/AFL/AT) documented by 12-lead ECG, surface ECG rhythm strips, 24-hour ambulatory ECG (Holter) monitor, or on ICM between days 91 and 365 following AAD initiation or AF ablation.

Secondary outcomes are listed in Table 4 of the Supplementary Appendix. These outcomes focus on AF progression ("time to first episode of persistent AF (>7 days)") and AF burden ("% time in AF"), including examining the relationship between AF burden and healthcare utilisation, and the relationship between AF burden and HRQOL.

ELIGIBILITY:
Inclusion Criteria:

• Non-permanent AF documented on a 12 lead ECG, Trans Telephonic Monitoring (TTM) or Holter monitor within the last 24 months, defined as:

i) Low Burden Paroxysmal - ≥2 episodes of AF over the past 12 months; Episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.

ii) High Burden Paroxysmal - ≥4 episodes of AF over the past 6 months, with ≥2 episodes >6 hours in duration; Episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.

iii) Early Persistent - ≥2 episodes of AF over the past 12 months; Episodes are successfully terminated via cardioversion within 7 days of onset.

* Age of 18 years or older on the date of consent
* Candidate for ablation based on AF that is symptomatic
* Informed Consent

Exclusion Criteria:

* Regular (daily) use of a class 1 or 3 antiarrhythmic drug (pill-in-the-pocket AAD use is permitted) at sufficient therapeutic doses according to guidelines (flecainide >50 mg BID, sotalol >80 mg BID, propafenone >150 mg BID
* Previous left atrial (LA) ablation or LA surgery
* AF due to reversible cause (e.g. hyperthyroidism, cardiothoracic surgery)
* Active Intracardiac Thrombus
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Left atrial anteroposterior diameter greater than 5.5 cm by transthoracic echocardiography
* Cardiac valve prosthesis
* Clinically significant (moderately-severe, or severe) mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* NYHA class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) less than 35%
* Hypertrophic cardiomyopathy (septal or posterior wall thickness >1.5 cm)
* Significant Chronic Kidney Disease (CKD - eGFR <30 µMol/L)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (strokes or TIAs) during the six-month interval preceding the consent date
* Pregnancy
* Life expectancy less than one (1) year
* Currently participating or anticipated to participate in any other clinical trial of a drug, device or biologic that has the potential to interfere with the results of this study
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2017-01; Primary Completion 2022-09 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence of symptomatic or asymptomatic Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia | Time to first recurrence between days 91 and 365 following treatment initiation
  The single procedure success (in the absence of AAD) is defined as the time to first recurrence of symptomatic** or asymptomatic AF, atrial flutter, or atrial tachycardia (AF/AFL/AT) documented by 12-lead ECG, surface ECG rhythm strips, ambulatory ECG monitor, or on implantable loop recorder and lasting 120 seconds or longer as adjudicated by a blinded group of investigators between days 91 and 365 post randomization.

SECONDARY OUTCOMES:
Time to recurrence of symptomatic AF/AFL/AT | Time to first recurrence between day 0 and 365 post Ablation
  Time to first recurrence of symptomatic documented AF/AFL/AT between days 91 and 365 after ablation or a repeat ablation procedure between days 0 and 365 post ablation.
Total arrhythmia burden | From 91 to 365 days following treatment initiation
  Total arrhythmia burden (daily AF burden - hours/day; overall AF burden - % time in AF)
Total arrhythmia burden | From 91 days following treatment initiation to final follow-up (~36 months)
  Total arrhythmia burden (daily AF burden - hours/day; overall AF burden - % time in AF)
Major complications of ablation, or significant adverse drug events (death, ventricular pro-arrhythmia, syncope, hypotension requiring hospitalisation, pacemaker insertion). | Acute peri-procedural complications will be defined as occurring within 30 days of ablation, with delayed complications occurring 31-365 days after ablation.
  Events include events death, ventricular pro-arrhythmia, syncope, hypotension requiring hospitalisation, pacemaker insertion).
Economic Evaluation | to end of follow up at 36 months for each patient
  Incremental cost effectiveness ratio (ICER) for ony QALY gain
Health-related quality of life | Baseline, 12, 24, and 36 months following treatment initiation
  Disease-specific AFEQT score, Generic EQ-5D score
Symptom Status | Baseline, 12, 24, and 36 months following treatment initiation
  Freedom from symptoms attributable to atrial fibrillation
Healthcare utilisation | 12 and 36 months following treatment initiation
  Emergency visit, cardioversion, and hospitalization >24 hours in a healthcare facility
Non-Protocol Ablation Procedure | Treatment initiation to 365 days following treatment initiation
  Repeat ablation procedures in those randomized to first line catheter ablation, or any ablation procedure performed in patients randomized to AAD therapy
Non-Protocol Ablation Procedure | Treatment initiation to final follow-up (~36 months)
  Repeat ablation procedures in those randomized to first line catheter ablation, or any ablation procedure performed in patients randomized to AAD therapy
Safety Outcomes related to Ablation or AAD therapy | Treatment initiation to final follow-up (~36 months)
  Major complications of ablation, or significant adverse drug events (death, ventricular pro-arrhythmia, syncope, hypotension, pacemaker insertion).

OTHER OUTCOMES:
Time to first episode of persistent atrial tachyarrhythmia | From 91 days following treatment initiation to final follow-up (~36 months; Primary outcome of extended-follow-up study)
  Time to first occurrence of symptomatic or asymptomatic persistent atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL], or atrial tachycardia [AT]), as defined as the first occurrence of a continuous atrial tachyarrhythmia episode lasting ≥ 7 days in duration, or lasting 48 hours to 7 days in duration but requiring cardioversion for termination, as documented by implantable loop recorder.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Andrade, M.D., Principal Investigator — University of British Columbia
Locations (18):
- Canada (18):
  - Libin CV Calgary, Calgary, Alberta
  - Royal Alexandra, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Queen Elizabeth II, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Mary's Kitchener, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Rouge Valley Health System, Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
  - Le Centre hospitalier universitaire de Sherbrooke CHUS, Sherbrooke, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Andrade JG, Moss JWE, Kuniss M, Sadri H, Wazni O, Sale A, Ismyrloglou E, Chierchia GB, Kaplon R, Mealing S, Bainbridge J, Bromilow T, Lane E, Khaykin Y. The Cost-Effectiveness of First-Line Cryoablation vs First-Line Antiarrhythmic Drugs in Canadian Patients With Paroxysmal Atrial Fibrillation. Can J Cardiol. 2024 Apr;40(4):576-584. doi: 10.1016/j.cjca.2023.11.019. Epub 2023 Nov 23. PMID 38007219
- [Derived] Leon-Acuna IG, Suzuki T. Progression of Atrial Fibrillation after Cryoablation. N Engl J Med. 2023 Apr 6;388(14):1339-1340. doi: 10.1056/NEJMc2301604. No abstract available. PMID 37018501
- [Derived] Andrade JG, Deyell MW, Macle L, Wells GA, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Cadrin-Tourigny J, Kochhauser S, Verma A; EARLY-AF Investigators. Progression of Atrial Fibrillation after Cryoablation or Drug Therapy. N Engl J Med. 2023 Jan 12;388(2):105-116. doi: 10.1056/NEJMoa2212540. Epub 2022 Nov 7. PMID 36342178
- [Derived] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159
- [Derived] Andrade JG, Champagne J, Deyell MW, Essebag V, Lauck S, Morillo C, Sapp J, Skanes A, Theoret-Patrick P, Wells GA, Verma A; EARLY-AF Study Investigators. A randomized clinical trial of early invasive intervention for atrial fibrillation (EARLY-AF) - methods and rationale. Am Heart J. 2018 Dec;206:94-104. doi: 10.1016/j.ahj.2018.05.020. Epub 2018 Oct 18. PMID 30342299